CLINICAL TRIAL: NCT00780325
Title: A Single Center, Double-blind, Placebo-controlled Phase I Single-dose Cross-over Study in Healthy Subjects to Investigate the Inhibitory Effect of CG100649, Celecoxib, Naproxen, and Acetazolamide on the Activity of Cyclooxygenases (COX-1, COX-2) and Carbonic Anhydrases (CA-I, CA-II)
Brief Title: Effects of Dual Cyclooxygenase-2 and Carbonic Anhydrase Inhibition
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A total of three parts were planned for this study. The sponsor funded only Part 1, so that neither Part 2 nor Part 3 of this study has been conducted.
Sponsor: University of Pennsylvania (Other)
Collaborators: CrystalGenomics, Inc. (Industry)
Responsible Party: Principal Investigator, Carsten Skarke, MD, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 807821
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
Keywords: Cyclooxygenase-2; Carbonic anhydrase; Eicosanoids; Healthy volunteers
MeSH Terms: interventions — CG100649; Celecoxib; Naproxen; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): CG100649, single oral dose of 2 mg
  Interventions: Drug: CG100649 (2 mg)
- 2 (Experimental): CG100649, single oral dose of 8 mg
  Interventions: Drug: CG100649 (8 mg)
- 3 (Active Comparator): Celecoxib, single oral dose of 200 mg
  Interventions: Drug: Celecoxib
- 4 (Active Comparator): Naproxen, single oral dose of 500 mg
  Interventions: Drug: Naproxen
- 5 (Active Comparator): Acetazolamide, single oral dose of 250 mg
  Interventions: Drug: Acetazolamide
- 6 (Placebo Comparator): Placebo, single oral administration
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: CG100649 (2 mg) — CG100649 capsules: 2 mg, single oral administration (Part 1); CG100649 capsules: dose to be determined, single oral administration (the single CG100649 dose level used in Part 3 will be determined by part 1 and 2).
  Arms: 1
Drug: Celecoxib — Celecoxib (Celebrex®) capsules: 200 mg; single oral administration (Part 1 and 3)
  Other Names: Celebrex®
  Arms: 3
Drug: Placebo capsules — Placebo capsules: 198 mg silicified microcrystalline cellulose + 2 mg talc, multiple oral administrations (Part 1 and 3)
  Other Names: silicified microcrystalline cellulose
  Arms: 6
Drug: Naproxen — Naproxen (Naprosyn®) tablets: 500 mg, single oral administration (Part 3)
  Other Names: Naprosyn®)
  Arms: 4
Drug: Acetazolamide — Acetazolamide (generic, immediate release) tablets: 250 mg, single oral administration (Part 3)
  Other Names: generic Acetazolamide
  Arms: 5
Drug: CG100649 (8 mg) — CG100649 capsules: 8 mg, single oral administration (Part 1); CG100649 capsules: dose to be determined, single oral administration (the single CG100649 dose level used in Part 3 will be determined by part 1 and 2).
  Arms: 2

SUMMARY:
Cyclooxygenase-2 (COX-2) inhibitors have become a common analgesic treatment option for patients with arthritis. However, long-term treatment has been associated with increased cardiovascular risk. With the past withdrawals and rejections of approval for COX-2 inhibitors the treatment options are now very limited.

This translates for example to about 10 million osteoarthritis patients in the US who cannot receive COX-2 inhibitors because of concomitant hypertension. And this exemplifies the unmet medical need to develop and offer safe treatment options for this particular patient population.

This trial investigates pharmacodynamic aspects of CG100649 which is being developed as a novel COX-2 inhibitor. Preclinical data show a dual mechanism of action, which consists of the inhibition of the two enzymes COX-2 and carbonic anhydrase-I/-II (CA-I/II) and through which the cardiovascular risk of COX-2 inhibition might be attenuated.

DETAILED DESCRIPTION:
Part 1 and 2 (staged analysis): Single dose of study drugs [celecoxib, placebo] followed by 3 days of blood draws as Period I; then after a wash-out phase, single dose of study drugs [CG100649 2mg and 8mg, celecoxib 200mg, placebo], followed by blood draws on 6 days and bi-weekly urine collections for 8 weeks.

Part 3: Five-way cross-over of single doses of study drugs with a CG100649 single dose level as determined by part 1 and 2, celecoxib 200mg, naproxen 500mg, acetazolamide 250mg and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old, able and willing to provide written informed consent to participate in the study;
2. Subjects must be in generally good health as determined by pre-study medical history, physical examination, clinical laboratory tests and 12-lead electrocardiogram (ECG);
3. Body mass index (BMI) 19-32 kg/m2;
4. Normal blood pressure (BP) [systolic BP 90-140 mmHg, diastolic BP 50-90 mmHg] and heart rate (HR) [resting HR 45-90 bpm] without medication;
5. Clinical chemistry profile including electrolytes, alkaline phosphatase (ALK), lactate dehydrogenase (LDH), creatine phosphokinase (CPK), creatinine, and urea must be within the normal range without medication; screening liver enzymes may be up to 1.5x normal range; screening CPK must be within 2x normal range without medication;
6. Urinalysis including urinary creatinine must be within normal limits (trace findings and minor deviations are acceptable per the clinical decision of the Principal Investigator);
7. Subjects must be non-smokers and non-drinkers or willing to abstain from smoking, alcohol, caffeine and high-fat foods for the duration of study;
8. Subjects must be able to read, understand and follow the study instructions;
9. Subjects and their sexual partners must agree to use double barrier contraception during the study period and for 2 months afterward or provide proof of surgical sterility. Double barrier contraception may include, but is not limited to, using a male condom with spermicide; having a female sexual partner who agrees to use an IUD with spermicide, a female condom with spermicide, a diaphragm with spermicide, a cervical cap with spermicide; or having a sterile sexual partner. Female subjects must be non-pregnant, non-lactating, and either postmenopausal for at least 1 year, surgically sterile for at least 3 months, or willing to use double barrier contraception from 28 days prior to study enrollment and/or their last confirmed menstrual period (whichever is longer) until 2 months after final clinic visit. For all females, the pregnancy test result must be negative at Screening;
10. Subjects must tolerate the insertion of an intravenous line of the size ≥ 20 gauge for the drug administration study days.

Exclusion Criteria:

1. Use of any non-study medication(s) including low dose aspirin for cardiovascular prophylaxis within 2 weeks prior and 2 weeks after receipt of each dose of study drug;
2. Use of chemotherapy agents or history of cancer, other than non-metastatic skin cancer that has been completely excised, within five (5) years prior to the screening visit;
3. History of bacterial or viral infection requiring treatment with antibiotics or antivirals within 3 months of study;
4. Presence or history of peripheral edema within the past 5 years;
5. History of congestive heart failure;
6. Use of drugs which are P450 3A4 inducers or inhibitors within the past 30 days (e.g. alprazolam, chlorpheniramine, cimetidine, fluoxetine, haloperidol, ketoconazole, itraconazole, erythromycin, clarithromycin, sildenafil, simvastatin, St. John's Wort);
7. Use of prescribed systemic or topical medications or any dietary aids or foods that are known to modulate drug metabolizing enzymes (e.g. grapefruit juice) within 14 days of dose administration;
8. Difficulty in swallowing oral medications;
9. History of seizure disorder;
10. Serious psychosocial co-morbidities;
11. Cognitive or psychiatric disorders, or any other condition that could interfere with compliance with study procedures and/or confinement in a clinical study unit for 2 days or longer;
12. History of drug or alcohol abuse within one year prior to screening;
13. Use of any other investigational drug within 1 month prior to enrollment;
14. Use of any prescription drugs within 1 month prior to enrollment;
15. Use of over the counter medication excluding routine vitamins, but including mega-dose vitamin therapy, within one week of enrollment;
16. Donation and/or receipt of any blood or blood products within 3 months prior to enrollment;
17. Active gastrointestinal, renal, hepatic, or coagulant disorder within 1 month prior to enrollment;
18. Esophageal or gastroduodenal ulceration within 1 month prior to enrollment;
19. Hypersensitivity to NSAIDs, sulfonamides, COX-2 inhibitors, or carbonic anhydrase inhibitors;
20. Known allergy or hypersensitivity to sulfa drugs;
21. Family history of significant cardiac disease (i.e. sudden death in first degree relative; myocardial infarction prior to 50 years old);
22. Occult blood in stool (fecal occult blood test).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Study compound-induced changes on the TxB2 formation in plasma and the formation of prostacyclin metabolite (PGI-M) in urine (Part 1) | Hours and days
Study compound-induced changes on urinary eicosanoid metabolites (Part 2) | Hours and days.
The study compound's biochemical selectivity for COX-2 (Part 3) | Hours and days.

SECONDARY OUTCOMES:
Study compound-induced changes on the urinary metabolites PGE-M and TxB-M; on the cyclooxygenase-2 dependent PGE2 production in ex vivo LPS-stimulated monocytes and on the carbonic anhydrase-I and II function; Biochemical selectivity for COX-2 (Part 1) | Hours and days
Inhibition of carbonic anhydrase and relationship to drug concentrations; Study compound-induced changes on serum TxB2, on PGE2 formation in LPS-stimulated monocytes, on PGI-M, PGE-M, TxB-M and PGD-M levels and on platelet aggregation (Part 3) | Hours and days

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine; Carsten C Skarke, MD, Principal Investigator — Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine; William K Schmidt, PhD, Study Director — CrystalGenomics, Inc.
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Skarke C, Alamuddin N, Lawson JA, Cen L, Propert KJ, Fitzgerald GA. Comparative impact on prostanoid biosynthesis of celecoxib and the novel nonsteroidal anti-inflammatory drug CG100649. Clin Pharmacol Ther. 2012 Jun;91(6):986-93. doi: 10.1038/clpt.2012.3. Epub 2012 Jan 25. PMID 22278334
- [Result] Hirankarn S, Barrett JS, Alamuddin N, FitzGerald GA, Skarke C. GCG100649, A Novel Cyclooxygenase-2 Inhibitor, Exhibits a Drug Disposition Profile in Healthy Volunteers Compatible With High Affinity to Carbonic Anhydrase-I/II: Preliminary Dose-Exposure Relationships to Define Clinical Development Strategies. Clin Pharmacol Drug Dev. 2013 Oct;2(4):379-86. doi: 10.1002/cpdd.47. Epub 2013 Jul 25. PMID 27121942